CLINICAL TRIAL: NCT03616184
Title: A Single Arm, Open Label, Phase II Study of Ruxolitinib in Sclerotic Chronic Graft-Versus-Host Disease After Failure of Systemic Glucocorticoids
Brief Title: Study of Ruxolitinib in Sclerotic Chronic Graft-Versus-Host Disease After Failure of Systemic Glucocorticoids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0333-18-FB
Record Dates: First submitted 2018-07-29; First posted 2018-08-06 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Graft-versus-host-disease (GVHD)
MeSH Terms: conditions — Graft vs Host Disease | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib (Experimental): Patients will receive oral ruxolitinib at a dose of 10 mg twice daily.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Patients with sclerotic chronic graft-versus-host disease (GVHD) will receive oral ruxolitinib at a dose of 10 mg twice daily. Doses may not exceed 10 mg twice daily. Ruxolitinib will be continued for 6 months. Patients who continue to have stable disease, mixed responses or partial/complete responses at the end of 6 months may continue the drug for a total of 12 months.

SUMMARY:
The primary objective of the study is to examine the efficacy of ruxolitinib in patients with sclerotic chronic graft-versus-host disease (GVHD).

DETAILED DESCRIPTION:
Chronic graft-versus-host-disease (GVHD) is a major complication of allogeneic hematopoietic cell transplant that impairs quality of life, and is associated with significant morbidity and mortality. Management of chronic GVHD with prednisone is associated with an overall response rate of approximately 60%, and a complete response rate of approximately 30% but sclerotic features do not respond as well. Based on the biology of chronic GVHD and available preliminary evidence, the investigators hypothesize that ruxolitinib will be effective in the management of sclerotic chronic GVHD. The study is an open label, phase II multicenter trial designed to evaluate the efficacy of ruxolitinib as a salvage treatment for patients with sclerotic GVHD (sclerosis or fasciitis). The primary objective is to determine the proportion of patients with response rate (complete and partial responses) in skin and/or joint, as determined by 2014 NIH (National Institutes of Health) consensus criteria, at 6 months of therapy with ruxolitinib. Eligibility criteria includes adult patients with chronic GVHD and skin, joint and/or fascia sclerosis, who have received systemic corticosteroids for >12 months and at least one additional line of therapy OR systemic corticosteroids and at least two additional lines of therapy for chronic GVHD. A sample size of 47 patients (43 evaluable patients and estimated 10% dropout) will allow an α of 0.044 and a power of 84% to test the null hypothesis response rate of 25% compared to an alternative of 45%. Subjects will receive ruxolitinib for 6 months for the treatment of sclerotic chronic GVHD. Subjects will be evaluated for GVHD status as well as non-relapse mortality, relapse of underlying malignancy and quality of life/functional status. Plasma cytokine levels and T/Natural Killer (NK) cell subset in peripheral blood will be measured at various time points. The response rate will be reported as a proportion and 95% exact confidence interval. If positive, the trial results will support other ongoing studies to establish the role of ruxolitinib in chronic GVHD in general and specifically in sclerotic chronic GVHD.

ELIGIBILITY:
Inclusion Criteria:

1. Sclerotic chronic GVHD (classic chronic or overlap syndrome) that meets 2014 NIH Consensus Criteria. Eligible patients will have superficial or deep skin sclerosis, fasciitis or joint contractures.
2. The subject must have received the following therapy for chronic GVHD (not necessarily for sclerotic manifestations): A - Systemic corticosteroids for >12 months and at least one additional line of systemic therapy OR B - Systemic corticosteroids and at least two additional lines of systemic therapy. For the purpose of this study, fluticasone, azithromycin and montelukast ("FAM") therapy for lung GVHD will be considered a topical therapy. Investigators are encouraged but not mandated to use ibrutinib for appropriate patients prior to enrollment in this trial.
3. Adults, Age ≥18 years (state of Nebraska, Age ≥19 years)
4. Karnofsky performance status ≥60% at the time of enrollment
5. All allogeneic donor sources and all conditioning regimens are allowed.
6. Absolute neutrophil count (ANC) greater than 1000/µL, and platelet count ³50,000/µL without the use of growth factors or platelet transfusion.
7. Able to take orally-administered medication.
8. Female patient of reproductive potential must have a negative serum or urine pregnancy test ≤7 days prior to starting the study drug. Women are considered NOT to have reproductive potential if they have had 12 months of amenorrhea with an appropriate clinical profile (i.e. ≥51 years, history of vasomotor symptoms, OR supportive hormone levels such as low estrogen and high follicle-stimulating hormone levels), OR surgical sterilization.
9. Male and female patients of reproductive potential must be willing to avoid pregnancy or fathering children from enrollment to one month after the end of study treatment. This will require either a total abstinence, OR exclusively non-heterosexual activity (when this is in line with the preferred and usual lifestyle of the subject), OR two methods of contraception (male or female condom with or without a spermicidal agent, diaphragm or cervical cap with spermicide, or hormonal based contraception including intrauterine device).
10. Life expectancy greater than 6 months
11. Written informed consent to participate in the study.

Exclusion Criteria:

1. Fibrosis of internal organs such as gut, liver or lung as the sole manifestation of sclerosis.
2. Fluconazole at a dose more than 200 mg daily. Patients should stop fluconazole or lower dose to less than or equal to 200 mg daily before starting ruxolitinib.
3. Current evidence of malignancy after allogeneic transplant.
4. History of progressive multifocal leuko-encephalopathy (PML)
5. Active uncontrolled bacterial, fungal, parasitic, or viral infection. Infections are considered controlled if appropriate therapy has been instituted and, at the time of screening, no signs of infection progression are present. Progression of infection is defined as hemodynamic instability attributable to sepsis, new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection
6. Presence of known HIV infection, active hepatitis B or C infection.
7. Active tuberculosis infection that developed after allogeneic hematopoietic cell transplant (HCT)
8. Total bilirubin 1.5 ´ the upper limit of the normal range
9. Creatinine clearance <30 mL/min
10. 10. Presence of uncontrolled cardiopulmonary conditions such as ongoing cardiac arrhythmias, unstable angina or myocardial infarction, uncontrolled hypertension (e.g. blood pressure higher than 150/90 for patients 60 years or older, or higher than 140/90 for patients younger than 60 years, or those with diabetes and chronic kidney disease), New York Heart Association class III/IV congestive heart failure, or requirement of supplemental oxygen at rest or having a resting O2 saturation <90% by pulse oximetry.
11. Any other condition that is judged by the physician to potentially interfere with compliance to the study protocol or pose a significant risk to the patient.
12. Pregnancy, breastfeeding or planning to be pregnant.
13. Exposure to Janus kinase inhibitors (JAK) inhibitor therapy for any indication after allogeneic transplant
14. Initiation of a new systemic immunosuppressant for management of chronic GVHD within 8 weeks prior to enrollment. However, patients who develop disease progression can enroll as early as 4 weeks after initiation of a new systemic immunosuppressant. Also, patients who are unable to tolerate current therapy can enroll any time after initiation of a new systemic immunosuppressant, as long as the "new" immunosuppressant is stopped in these cases prior to initiation of ruxolitinib. Initiation of any new topical therapy (including FAM or intra-oral narrow-band UVB phototherapy) and changes in dose of existing immunosuppressive agents such as corticosteroids, sirolimus, calcineurin inhibitors or other agents are acceptable at any time prior to enrollment. The use of immunosuppressants for short term period, for example 7 days, for indications other than GVHD will be acceptable.
15. Treatment with any other investigational agent, device, or procedure, within 21 days (or 5 half-lives, whichever is greater)
16. Known allergies, hypersensitivity, or intolerance to any of the study medications, excipients, or similar compounds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2022-01-22 (Actual); Study Completion 2023-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vijaya Bhatt, MD, Principal Investigator — University of Nebraska
Locations (5):
- United States (5):
  - Moffitt Cancer Center, Tampa, Florida
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhatt VR, Shostrom VK, Choe HK, Hamilton BK, Gundabolu K, Maness LJ, Kumar V, Mahato RI, Smith LM, Nishihori T, Lee SJ. A Multicenter Phase II Trial of Ruxolitinib for Treatment of Corticosteroid Refractory Sclerotic Chronic Graft-Versus-Host Disease. J Clin Oncol. 2024 Nov 20;42(33):3977-3985. doi: 10.1200/JCO.24.00205. Epub 2024 Aug 16. PMID 39151112

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ruxolitinib
Started | 47
Completed | 34
Not Completed | 13

BASELINE CHARACTERISTICS:
Population: 49 patients were consented to the study, and 2 were screen fails. 47 patients received at least one dose of Ruxolitnib and were included in safety analyses.
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 47
Age, Continuous [Median (Full Range); unit: Years] | 62 [23 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 43
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete and Partial Responses in Skin and/or Joint
Description: The primary endpoint of the study was complete or partial response in skin and/or joint defined according to the 2014 NIH cGVHD Consensus Criteria. Partial response for skin would be a decrease in NIH Skin Score by 1 or more points. Partial response in joint would be a decrease in NIH Joint and Fascia Score by 1 or more points or increase in P-ROM score by 1 point for any site.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 34
percentage of participants | 49

2. Secondary Outcome: Percentage of Participants With Complete or Partial Responses Overall
Description: As determined by 2014 NIH Criteria which is a clinician overall severity score of 0 for complete response and clinician overall severity score decreased by 2 or more points on a 0-10 scale for partial response.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 34
percentage of participants | 47

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse Events were monitored/assessed/classified without regard to the specific Adverse Event Term.
Arm/Group | Ruxolitinib
All-Cause Mortality (participants affected / at risk) | 4/47
Serious Adverse Events (participants affected / at risk) | 13/47
Other Adverse Events (participants affected / at risk) | 29/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib (N=47)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Chest pain-cardiac (Cardiac disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Infections and infestations (Infections and infestations) | 1 (2)
Investigations (Investigations) | 4 (5)
Lung Infection (Infections and infestations) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sudden death NOS (General disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib (N=47)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 5 (8)
Dizziness (Nervous system disorders) | 3 (3)
Dry Eye (Eye disorders) | 3 (3)
Fatigue (General disorders) | 7 (8)
Hypertension (Vascular disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 8 (9)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (3)
Upper respiratory infection (Infections and infestations) | 8 (14)
Vomiting (Gastrointestinal disorders) | 6 (6)
weight gain (Investigations) | 5 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/84/NCT03616184/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/84/NCT03616184/ICF_000.pdf